CLINICAL TRIAL: NCT01076049
Title: Evaluation of a Novel Solution, IrriSept, a New Delivery System, Containing a Long-acting Antimicrobial Agent for Irrigation of Skin and Soft Tissue Infections, in the Form of an Abscess in the Emergency Department: a Pilot Study
Brief Title: The Effect of Irrisept for Irrigation of Skin and Soft Tissue Infections (Irrisept USF Study)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Suboptimal Recruitment
Sponsor: Irrimax Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 108527
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Results first posted 2021-07-28 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Skin and Soft Tissue Infections; Abscess
MeSH Terms: conditions — Soft Tissue Infections; Abscess

STUDY DESIGN:
Intervention Model Description: The randomization methodology was controlled by a biostatistician at the site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care (SoC) (Active Comparator): For subjects randomized to the control group, the preferred irrigation solution was chosen by the site's emergency department physician(s).
  Interventions: Device: Standard of Care (SoC)
- Irrisept (Active Comparator): For subjects randomized to the investigational group, Irrisept was used.
  Interventions: Device: Irrisept Delivery System

INTERVENTIONS:
Device: Standard of Care (SoC) — The preferred irrigation solution and method was chosen by the site's emergency department physician(s) and could vary between subjects. The type of SoC was recorded in the source document and the same solution and irrigation method were used during the initial treatment and 48-hour follow-up visits.
  Arms: Standard of Care (SoC)
Device: Irrisept Delivery System — Irrisept is a manual, self-contained irrigation device capable of producing 7-8 psi of pressure for effective wound cleansing and irrigation. Irrisept contents include the Chlorhexidine Gluconate (CHG) solution, a 450 mL bottle, and Irriprobe applicator or an abscess irrigation tip. The bottle design allows users to control the pressure of the solution through manual bottle compression.
  Irrisept was recorded in the source document and used during the initial treatment and 48-hour follow-up visits.
  Other Names: Irrisept
  Arms: Irrisept

SUMMARY:
The purpose of this study was to determine whether Irrisept can effectively prevent the progression of skin and soft tissue infections (SSTIs) as compared to treatment by the current Standard of Care.

DETAILED DESCRIPTION:
After being informed about the trial and potential risks, subjects completed an informed consent form prior to participation. After eligibility criteria was verified, an initial wound assessment examination was performed. Subjects were then randomized to the Irrisept or Standard of Care treatment group. Forty-eight hours later, wound progression and signs of infection were assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80
2. Skin and soft tissue infections (SSTIs), in the form of an abscess, which will require incision and drainage.
3. Patient able to provide an informed consent.
4. Patient volunteers to participate.

Exclusion Criteria:

1. Wound was caused by human or animal bite.
2. Wound is a blunt crush injury or has tendon, bone, or joint involvement.
3. Diabetic foot infection.
4. Anticipated incision size less than 5mm.
5. Abscess extends to the muscle layer.
6. Admission to hospital for any reason, including IV antibiotics.
7. Clinical signs of systemic infection on initial patient encounter.
8. Prior history of allergy or hypersensitivity to CHG.
9. Neutropenic (known ANC<500/mm3), HIV (known CD4<50), or other severely immunocompromised state (e.g., receiving chemotherapy).
10. Patient is diagnosed with systemic lupus erythematosus or other immunological disease.
11. Currently in police custody.
12. Patient withdraws from participation.
13. Patient unable or unwilling to give informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wein, MD, Principal Investigator — Tampa General Hospital, University South Florida
Locations (1):
- Tampa General Hospital - University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 2010 to December 2011, patients with skin and soft tissue infections were recruited from the Tampa General Hospital, University of South Florida emergency department.
Pre-assignment Details: A total of 114 subjects consented to the study. Of these, 107 subjects were randomized as six (6) failed screening and one (1) subject had no randomization information available, but still completed the study. In total, 98 subjects completed the study. Of those 98 subjects, 52 subjects were enrolled in the Irrisept arm and 45 subjects were enrolled in the SoC control arm. There are records of an additional subject completing the study, but no randomization information was available.
Groups:
- Standard of Care (SoC): The type of irrigation solution and method used as SoC was determined by the participating emergency department physician. The SoC method was used at the initial and 48-hour follow-up visit.
- Irrisept Delivery System: Irrisept was recorded in the source document and used during the initial treatment and 48-hour follow-up visits.
  Irrisept is a manual, self-contained irrigation device capable of producing 7-8 psi of pressure for effective wound cleansing and irrigation. Irrisept contents include the Chlorhexidine Gluconate (CHG) solution, a 450 mL bottle, and Irriprobe applicator or an abscess irrigation tip. The bottle design allows users to control the pressure of the solution through manual bottle compression.
- Randomization Unknown: The randomization group (SoC or Irrisept) is unknown for 1 subject.
Period: Overall Study
Arm/Group | Standard of Care (SoC) | Irrisept Delivery System | Randomization Unknown
Started | 52 | 55 | 1
Completed | 45 | 52 | 1
Not Completed | 7 | 3 | 0

BASELINE CHARACTERISTICS:
Population: A total of 114 subjects were consented. There were 6 screen failures. There were 107 subjects randomized (55 to Irrisept and 52 to SoC). One (1) subject had no randomization information available. There were 52 Irrisept and 45 SoC subjects that completed the trial. For one SoC subject, the gender is unknown.
Groups:
- Irrisept Device System: For subjects randomized to the investigational group, Irrisept was used.
  Irrisept Delivery System: Irrisept is a manual, self-contained irrigation device capable of producing 7-8 psi of pressure for effective wound cleansing and irrigation. Irrisept contents include the Chlorhexidine Gluconate (CHG) solution, a 450 mL bottle, and Irriprobe applicator or an abscess irrigation tip. The bottle design allows users to control the pressure of the solution through manual bottle compression.
  Irrisept was recorded in the source document and used during the initial treatment and 48-hour follow-up visits.
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SoC) | Irrisept Device System | Randomization Unknown | Total
Number analyzed (Participants) | 45 | 52 | 1 | 98
Age, Customized [Count of Participants; unit: Participants]
  Subject Accounting | 45 | 52 | 1 | 98
Sex/Gender, Customized [Count of Participants; unit: Participants] — There were 52 Irrisept and 45 SoC subjects that completed the trial. For one SoC subject, the gender is unknown.
  Participants
    Gender: Female | 25 | 27 | 0 | 52
    Gender: Male | 19 | 25 | 1 | 45
    Gender: Unknown Gender | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race (Black) | 15 | 25 | 0 | 40
  Race (White) | 23 | 18 | 1 | 42
  Ethnicity (Hispanic) | 6 | 7 | 0 | 13
  Unknown Race/Ethnicity | 1 | 2 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 52 | 1 | 98

OUTCOME MEASURES:

1. Primary Outcome: Wound State at 48-Hour Follow-up Visit
Description: The primary endpoint was overall wound progression and signs of infection 48 hours post-treatment. This was measured via a blinded investigator's discretion and recorded as 'improved', 'no change', 'progression of signs or symptoms of infection', or 'immediate treatment required' if an infection had progressed to a certain extent.
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) | Irrisept Device System | Randomization Unknown
Number analyzed (Participants) | 45 | 52 | 1
Participants
  Improved Wound State at 48-Hour Follow-up | 40 | 47 | 0
  No Change Wound State at 48-Hour Follow-up | 1 | 1 | 0
  Progression Wound State at 48-Hour Follow-up | 3 | 2 | 0
  Immediate Treatment Required Wound State at 48-Hour Follow-up | 1 | 2 | 1

2. Secondary Outcome: Clinical Performance of Irrisept to the Current SoC
Description: The study tracked any instance of a subject's conditions worsening compared to their baseline measurements. This included a worsening in the size (length and width) and clinical signs (erythema, area, induration, tenderness, warm, pain, cellulitis and other) of the infection.
  While the protocol states the overall prevalence of Methicillin-resistant Staphylococcus Aureus (MRSA) colonization is the secondary objective, this information was not collected by the site. Therefore, worsening of clinical outcomes is considered the secondary objective.
Time Frame: 48 hours
Population: There were 45 SoC & 52 Irrisept subjects that completed the trial. Of these, 20 SoC & 16 Irrisept subjects showed clinical signs of infection worsening; 25 SoC & 36 Irrisept subjects did not show infection worsening signs. Worsening signs include changes in length, width, erythema, area, induration tenderness, warmth, pain, cellulitis and other. The total number of worsening signs for SoC subjects was 32. The total number of worsening signs for Irrisept subjects was 28.
Measure: Number; unit: Total Number of Worsening Outcomes
Units Other Than Participants: Total Number of Worsening Outcomes
Arm/Group | Standard of Care (SoC) | Irrisept Delivery System | Randomization Unknown
Number analyzed (Participants) | 45 | 52 | 1
Number analyzed (Total Number of Worsening Outcomes) | 32 | 28 | 1
Total Number of Worsening Outcomes
  Increased Length (cm) | 5 | 9 | 0
  Increased Width (cm) | 3 | 5 | 1
  Erythema | 4 | 0 | 0
  Area (cm2) | 1 | 3 | 0
  Induration | 6 | 2 | 0
  Tenderness | 2 | 2 | 0
  Warmth | 6 | 3 | 0
  Pain | 3 | 3 | 0
  Cellulitis | 0 | 0 | 0
  Other | 2 | 1 | 0
  No Signs of Infection Worsening | 25 | 36 | 0

3. Post Hoc Outcome: Worsening Events Causality
Description: Causality for each worsening event was determined by using the following categories: 'related', 'possibly related', 'unlikely related', or 'unrelated'.
Time Frame: 48 Hours
Population: Causality assessment categories for each worsening sign were related, possibly related, unlikely related, or unrelated. 45 SoC and 52 Irrisept subjects completed the trial. Of these, 20 SoC & 16 Irrisept subjects showed clinical signs of worsening; causality assessments were made for each worsening sign (ex: length, erythema, etc.). There were 32 and 28 total worsening signs for SoC & Irrisept subjects, respectively.
Measure: Count of Units; unit: Total Number of Worsening Outcomes
Units Other Than Participants: Total Number of Worsening Outcomes
Arm/Group | Standard of Care (SoC) | Irrisept Delivery System | Randomization Unknown
Number analyzed (Participants) | 45 | 52 | 1
Number analyzed (Total Number of Worsening Outcomes) | 32 | 28 | 1
Total Number of Worsening Outcomes
  Related Worsening Event | 0 | 0 | 0
  Possibly Related Worsening Event | 0 | 0 | 0
  Unlikely Related Worsening Event | 28 | 26 | 0
  Unrelated Worsening Event | 4 | 2 | 1

ADVERSE EVENTS:
Time Frame: The timeframe used for reporting adverse events was from the time of informed consent until subject termination or completion (approximately 48 hours after the initial visit).
Description: Any change in the subjects' wound infection (i.e. any worsening of the secondary objective clinical outcomes) were considered adverse events. Causality assessments were provided. All-cause mortality and serious adverse events were not monitored nor assessed.
Groups:
- Randomization Unknown: There are records of an additional subject completing the study, but no randomization information was available.
Arm/Group | Standard of Care (SoC) | Irrisept Delivery System | Randomization Unknown
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 20/45 | 16/52 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SoC) (N=45) | Irrisept Delivery System (N=52) | Randomization Unknown (N=1)
Increased Length (Infections and infestations) | 5 (5) | 9 (9) | 0 (0) — Change in length, measured in cm.
Increased Width (Infections and infestations) | 3 (3) | 5 (5) | 1 (1) — Change in width, measured in cm.
Erythema (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Area (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) — Area, measured in cm2.
Induration (Infections and infestations) | 6 (6) | 2 (2) | 0 (0)
Tenderness (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Warmth (Infections and infestations) | 6 (6) | 3 (3) | 0 (0)
Pain (Infections and infestations) | 3 (3) | 3 (3) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)
Other (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-08-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT01076049/Prot_SAP_000.pdf